CLINICAL TRIAL: NCT00948194
Title: Investigation of the Effect of Nitric Oxide on Ischemic Reperfusion Injury During Extended Donor Criteria Liver Transplantation
Brief Title: Effect of Nitric Oxide (NO) on Ischemic/Reperfusion Injury During Extended Donor Criteria (EDC) Liver Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was terminated when the P.I. left the university.
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09-0137
Record Dates: First submitted 2009-07-24; First posted 2009-07-29 (Estimated); Results first posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Liver Transplantation; Ischemia/Reperfusion Injury; Oxidative Injury
Keywords: Extended Donor Criteria
MeSH Terms: conditions — Reperfusion Injury | interventions — Nitric Oxide; Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No nitric oxide (No Intervention): This arm will not receive nitric oxide, but will receive other standard inhaled anesthetics
- Nitric Oxide (Experimental): Will receive Nitric oxide and other standard inhaled anesthetics
  Interventions: Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitric Oxide — Inhalation - 40 ppm, at the initiation of anesthesia to the end of surgery
  Other Names: INOmax
  Arms: Nitric Oxide

SUMMARY:
In this study, the researchers propose to investigate the efficacy of inhaled nitric oxide to prevent ischemia-reperfusion (I/R) hepatocyte injury in patients who receive extended donor criteria(EDC)liver grafts based on changes in proteomic and metabolomic markers following revascularization of the donor graft.

In reviewing the literature, no uniform extended criteria donor classification exists. The characteristics most associated with liver graft failure appear to be cold ischemia time greater than 10 hours, warm ischemia time greater than 40 minutes, donor age > 55 years of age, donor hospitalization > 5 days, a donation after cardiac death (DCD) graft, and a split graft. The researchers will exclude warm ischemia time as this is impossible to predict prior to the transplantation. Any donor meeting at least one of the other criteria will be classified as an EDC donor.

Hypothesis 1: Inhaled nitric oxide will improve overall outcome of liver recipients after EDC liver transplantation

* Suppression of oxidative injury will improve graft function postoperatively as measured by International Normalized Ratio (INR) bilirubin, transaminases, and duration of hospital stay.

Hypothesis 2: The mechanisms of therapeutic efficacy of inhaled nitric oxide is based on reduction in post-reperfusion oxidative injury as readily measured by the detectable changes in the protein and metabolic profiles in plasma of patients treated with inhaled-NO

* Nuclear Magnetic Resonance (NMR)-based metabolic markers (xanthine end-products, lactate, and hepatic osmolytes) that are consistent with acute liver injury will be decreased in NO-treated recipients.
* Protein markers of reperfusion injury (argininosuccinate synthase (ASS) and estrogen sulfotransferase (EST-1) will be greater in the plasma of patients who are not treated with inhaled-NO
* Reduced oxidative injury will be reflected by a decrease in the number of mitochondrial peroxiredoxins isoforms and the number that are oxidized in NO-treated liver recipients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 69 years of age
* moderate to severe liver disease (MELD score 22 to 30)
* is receiving a extended donor criteria liver graft

Exclusion Criteria:

* undergoing multi-organ transplant
* 70 years or older
* diagnosed with hepatocarcinoma
* diagnosed with either hepatopulmonary syndrome or pulmonary hypertension
* pregnant

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J. Fiegel, M.D., Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Nitric Oxide | Nitric Oxide
Started | 6 | 7
Completed | 5 | 7
Not Completed | 1 | 0
Not completed — Blood drawn using incorrect test tube; sample invalid | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data was not collected one participant whose sample was invalid.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Nitric Oxide | Nitric Oxide | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 5 | 9
Diagnosis [Number; unit: participants]
  Cirrhosis | 5 | 3 | 8
  Hepatitis C | 4 | 4 | 8
  HCC | 2 | 4 | 6
  Hepatoma | 1 | 4 | 5
  Primary Sclerosing Cholangitis (PSC) | 0 | 1 | 1
  Fatty Liver (NASH) | 1 | 0 | 1
  Metabolic Disease (METDIS) - Alpha-1-Antitrypsin Deficiency (A-1-A) | 0 | 1 | 1
  Bone mets | 0 | 1 | 1
Model for End-Stage Liver Disease Score [Mean (Standard Deviation); unit: units on a scale] — The Model For End-Stage Liver Disease (MELD) score assesses the severity of patient liver disease. Possible scores range from 6 to 40, with higher scores indicating more severe liver disease and a worse outcome.
  units on a scale | 26.2 (5.42) | 27.14 (3.64) | 26.75 (4.5)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.59 (5.01) | 27.1 (5.83) | 26.89 (5.51)

OUTCOME MEASURES:

1. Primary Outcome: To Determine if Inhaled Nitric Oxide Has Beneficial Effects on Overall Outcome After Extended Criteria Donor (EDC) Liver Transplantation
Time Frame: 3 years
Population: The outcome measure data are unavailable. This study was terminated when the P.I. left the university. Research Administration and the study team have made numerous unsuccessful attempts to obtain the outcome measure data.
Arm/Group | No Nitric Oxide | Nitric Oxide
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Construct a Plasma Metabolic/Protein Profile of I/R Injury in Transplanted Livers
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | No Nitric Oxide | Nitric Oxide
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: To Examine the Effects of Nitric Oxide on Protein Synthesis and Metabolism Following Extended Criteria Donor Liver Transplantation
Time Frame: 3 years
Population: as for outcome 1
Arm/Group | No Nitric Oxide | Nitric Oxide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | No Nitric Oxide | Nitric Oxide
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7
Other Adverse Events (participants affected / at risk) | 0/5 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes